CLINICAL TRIAL: NCT03699722
Title: Developing a Women-Focused PrEP Intervention for HIV Prevention
Brief Title: A Women-Focused PrEP Intervention
Acronym: Just4Us
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: New York Blood Center (Other)
Responsible Party: Principal Investigator, Anne Teitelman, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R34MH108437-01A1 (NIH)
Record Dates: First submitted 2018-09-29; First posted 2018-10-09 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Behavior and Behavior Mechanisms; Information Literacy
Keywords: women; HIV; PrEP; intervention
MeSH Terms: conditions — Behavior | interventions — Educational Status; Exercise

STUDY DESIGN:
Intervention Model Description: At the baseline visit, participants will be randomly assigned to intervention or control conditions in a 3:1 ratio, stratified by site. Participants will remain in those assigned groups for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education + Activities (Experimental): 12 modules which include the following topics: introduction to the CN and intervention, video about PrEP, PrEP use in combination with other HIV, STI, and pregnancy prevention, identification and strategizing about beliefs regarding PrEP initiation, addressing perceived risk, strategizing about vulnerability factors that may interfere with PrEP uptake, skills building for PrEP uptake, and enhanced referral to a PrEP provider. Up to 4 follow-up phone calls to reinforce strategies. Text messaging for support PrEP adherence.
  Interventions: Behavioral: Education + Activities
- Information (Active Comparator): PrEP information brochures, frequently asked questions and questions to ask provider. Listing of local PrEP providers.
  Interventions: Behavioral: Information

INTERVENTIONS:
Behavioral: Education + Activities — Format:Video; discussion; information handouts; facilitated referral
  Arms: Education + Activities
Behavioral: Information — Format: Information handouts
  Arms: Information

SUMMARY:
Many women at high risk for acquiring HIV infection are not aware of preexposure prophylaxis (PrEP), an efficacious, self-administered, woman-controlled, HIV prevention product. The objective of this study is to evaluate the feasibility and acceptability of a theory-based intervention to promote PrEP uptake and adherence in a pilot trial among 80 women. The study will also measure intention to use PrEP and actual initiation of PrEP use. The investigators hypothesize that the intervention will be acceptable and feasible and that the intervention group will report higher levels of PrEP uptake, intention to use and adhere to PrEP, and other variables regarding PrEP uptake, comparing baseline, post-intervention and 3 month follow-up assessments.

DETAILED DESCRIPTION:
The HIV epidemic among women in the US is a major public health issue and many women at high risk for acquiring HIV infection are not aware of pre-exposure prophylaxis (PrEP), an efficacious, self-administered, woman-controlled, HIV prevention product. In 2014, the Centers for Disease Control and Prevention (CDC) and the American College of Obstetricians and Gynecologists (ACOG) issued guidelines for evaluating and prescribing PrEP for women at high risk for acquiring HIV. Yet, there are currently no interventions in the US to promote PrEP uptake among high risk women.

The objective of this study is to evaluate an intervention to promote PrEP uptake in two large metropolitan areas with local HIV rates that greatly exceed the national average but with different PrEP public policy and access landscapes. The investigators hypothesize that a theory-based, contextually relevant behavioral intervention combined with linkage to health care and social services, with text message support for adherence, would be feasible and acceptable and would improve PrEP uptake among high risk women.

Eligible women will be recruited primarily via face-to-face recruitment and respondent driven sampling. For respondent driven sampling, enrolled participants will be given three (3) coupons to be given to women in her social network who she thinks would be interested in joining the study. If the person referred attends a baseline visit, the referring participant will receive $10. Assessment of eligibility will be conducted by telephone or in-person. Participant initials and phone number will be recorded on the form. Eligible participants will be scheduled for a study visit at a day and time convenient for her. Study visits will be held at UPenn School of Nursing (Philadelphia) or the New York Blood Center Project Achieve office (NYC) or at a mutually agreeable location in the community that provides a private place for study procedures.

For the randomized trial, the investigators will conduct a study among 80 women to evaluate the feasibility and acceptability of the intervention. Each of the two study sites will enroll forty (40) women; thirty (30) participants will receive the theory-based, contextually tailored education and activities intervention and ten (10) participants will be randomized to the information only control group.

Prior to administering any study procedures women participants will participate in an informed consent process. During the informed consent process research staff will explained some participants will receive the education and activities intervention and some participants will receive information control group. After their questions are answered and participant signs the consent form, all participants will complete a computer-based baseline assessment and receive a rapid HIV test. All participants (control and intervention) will sign a release of information form authorizing the study team to contact the PrEP health care site for the minimal information needed to assess if PrEP was prescribed.

Randomization will be performed centrally by the project statistician, and implemented using opaque sealed envelopes. Envelopes will be numbered and shipped to each study site. Balance between arms will be maintained by use of randomly permutated blocks with unequal block sizes of 4 and 8 (to allow for the 3:1 randomization ratio), and with stratification by site (2 strata). At each site, a sealed envelope will be opened, in consecutive order, indicating study arm.

Upon completing the computer-based survey, participants randomized to the education and activities intervention arm will receive an individual tailored in-person session, conducted by a trained counselor/navigator (CN). Participants will also be asked to design simple personalized text messages for asking about PrEP initiation and PrEP adherence reminders once starting PrEP. Finally, the CN will also coordinate with the participant the best day and time to schedule her four (4) follow-up phone calls. During the phone calls, the CN will reinforce skills for PrEP uptake, review the action plan regarding identified vulnerability factors that could interfere with PrEP uptake and reinforce strategies to access referrals.

Participants randomized to the information only arm will meet with the counselor/navigator to review resources regarding PrEP and receive a list of providers/clinics prescribing PrEP.

After the session, participants will complete a post-session computer-bases survey to assess social-cognitive variables targeted in the intervention. Participants will also complete a Participant's Brief Satisfaction Questionnaire to provide feedback on the session.

All participants will be compensated $50.00 All participants enrolled will return to the study site for a three (3) month follow-up study visit to complete the computer-based survey and a questionnaire evaluating her experience navigating through the process to obtain provider appointment, medical assessment for PreP, prescription and taking PreP. Participants will be compensated $50.00 upon completing the three (3) month follow-up study visit.

ELIGIBILITY:
Inclusion Criteria:

* female at birth and identify as female
* aged 18-55;
* report unprotected vaginal or anal sex with a male partner OR any injection drug use in the past 6 months;
* live or have sex in a high risk area or are recruited into the study by someone who lives or has sex in a high risk area;
* understand and read English;
* not known to be HIV-infected;
* are willing to consider a daily pill with low rates of mild side effects to prevent HIV;
* have access to a mobile phone.
* report at least one of the following as 'yes' or 'do not know': current male partner who injects drugs or has sex with men; current male partner who is HIV infected; current male partner who was incarcerated in the last 6 months OR report at least one of the following as 'yes': shared injection equipment in last 6 months; in methadone, buprenorphine or suboxone treatment program in past 6 months; exchange sex for money, drugs, other goods in last 6 months; powder cocaine, crack use, methamphetamines, or ecstasy >1x/week in last 6 months; Chlamydia, syphilis, gonorrhea diagnosed or newly diagnosed genital herpes in last 6 months; alcohol abuse in last 6 months (defined as a score of 2 or higher on the CAGE36); has 3 or more male partners.

Exclusion Criteria:

* currently using PrEP

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 83 (Actual)
Dates: Start 2018-11-03 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
Intervention Fidelity | baseline session
  Evaluation of fidelity behavior for each module by site coordinator after listening to audio recordings of intervention sessions using a rating form with 90% evaluation items must be 4s or 5s on a 5-point Likert scale.
Participant Acceptability of intervention | baseline and 3 months
  At least 80% of participants report moderate or higher levels of acceptability: based on participants' indicating favorable responses indicated by 4s and 5s on a 5 point Likert scale on the Brief Satisfaction Questionnaire

SECONDARY OUTCOMES:
PrEP uptake behavior | 3 months
  PrEP uptake behavior (Preliminary Impact) as reported by self report at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Anne Teitelman, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We are happy to make our research findings readily available for research purposes to qualified individuals within the scientific community through individual requests directed to the Co-Principal Investigators and to share all published findings with the NIH. To protect confidentiality, qualitative data will be release in summary form. Findings from the study will be transmitted both to the scientific community through presentations at conferences and via journal articles and to interested community members through presentations. At each presentation and on each publication, contact information for additional information will be provided.

REFERENCES:
- [Derived] Teitelman AM, Tieu HV, Chittamuru D, Shaw PA, Nandi V, Davis A, Lipsky RK, Darlington CK, Fiore D, Koblin BA. A Randomized Controlled Pilot Study of Just4Us, a Counseling and Navigation Intervention to Promote Oral HIV Prophylaxis Uptake Among PrEP-Eligible Cisgender Women. AIDS Behav. 2023 Sep;27(9):2944-2958. doi: 10.1007/s10461-023-04017-z. Epub 2023 Mar 4. PMID 36869921
- [Derived] Teitelman AM, Koblin BA, Brawner BM, Davis A, Darlington C, Lipsky RK, Iwu E, Bond KT, Westover J, Fiore D, Tieu HV. Just4Us: Development of a Counselor-Navigator and Text Message Intervention to Promote PrEP Uptake Among Cisgender Women at Elevated Risk for HIV. J Assoc Nurses AIDS Care. 2021 Mar-Apr 01;32(2):188-204. doi: 10.1097/JNC.0000000000000233. PMID 33427767